CLINICAL TRIAL: NCT02439775
Title: Global Clinical Study of Renal Denervation With the Symplicity Spyral™ Multi-electrode Renal Denervation System in Patients With Uncontrolled Hypertension on Standard Medical Therapy (SPYRAL HTN-ON MED)
Brief Title: SPYRAL HTN-ON MED Study of Renal Denervation With the Symplicity Spyral™ Multi-electrode Renal Denervation System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPYRAL HTN-ON MED
Record Dates: First submitted 2015-04-28; First posted 2015-05-12 (Estimated); Results first posted 2023-09-15 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Hypertension; Vascular Diseases; Cardiovascular Diseases
Keywords: Uncontrolled hypertension; Renal denervation
MeSH Terms: conditions — Hypertension; Vascular Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (2):
- Renal Denervation (Experimental): Renal angiography and Renal Denervation (Symplicity Spyral™ multi-electrode renal denervation system)
  Interventions: Device: Symplicity Spyral™ multi-electrode renal denervation system
- Sham Procedure (Sham Comparator): Renal angiography
  Interventions: Procedure: Sham Procedure

INTERVENTIONS:
Device: Symplicity Spyral™ multi-electrode renal denervation system — After a renal angiography according to standard procedures, subjects remain blinded and are immediately treated with the renal denervation procedure after randomization.
  Other Names: Renal angiography; Renal Denervation
  Arms: Renal Denervation
Procedure: Sham Procedure — After a renal angiography according to standard procedures, subjects remain blinded and remain on the catheterization lab table for at least 20 minutes prior to introducer sheath removal.
  Other Names: Renal angiography
  Arms: Sham Procedure

SUMMARY:
The purpose of this study is to test the hypothesis that renal denervation decreases blood pressure and is safe when studied in the presence of up to three standard antihypertensive medications.

DETAILED DESCRIPTION:
The purpose of this study is to test the hypothesis that renal denervation is safe and reduces systolic blood pressure (SBP) in patients with uncontrolled hypertension on one, two, or three standard antihypertensive medications compared to a sham control in the same population. In this study, "uncontrolled hypertension" is defined as an office systolic blood pressure (SBP) ≥ 150 mmHg and <180 mmHg, an office Diastolic Blood Pressure (DBP) ≥90 mmHg and a 24-hour Ambulatory Blood Pressure Monitoring (ABPM) average SBP ≥140 mmHg to <170 mmHg, all of which are measured at Screening Visits. Data obtained will be used to confirm the effect of renal denervation on elevated blood pressure in patients on 1, 2 or 3 antihypertensive medications.

ELIGIBILITY:
Inclusion Criteria:

* Individual has office systolic blood pressure (SBP) ≥ 150 mmHg and <180 mmHg and a diastolic blood pressure (DBP) ≥ 90 mmHg when receiving a medication regimen of one, two, or three antihypertensive medication classes.
* Individual has 24-hour Ambulatory Blood Pressure Monitoring (ABPM) average SBP ≥ 140 mmHg and < 170 mmHg.

Exclusion Criteria:

* Individual lacks appropriate renal artery anatomy.
* Individual has estimated glomerular filtration rate (eGFR) of <45.
* Individual has type 1 diabetes mellitus or poorly-controlled type 2 diabetes mellitus.
* Individual has one or more episodes of orthostatic hypotension.
* Individual requires chronic oxygen support or mechanical ventilation other than nocturnal respiratory support for sleep apnea.
* Individual has primary pulmonary hypertension.
* Individual is pregnant, nursing or planning to become pregnant.
* Individual has frequent intermittent or chronic pain that results in treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) for two or more days per week over the month prior to enrollment
* Individual has stable or unstable angina within 3 months of enrollment, myocardial infarction within 3 months of enrollment; heart failure, cerebrovascular accident or transient ischemic attack, or atrial fibrillation at any time.
* Individual works night shifts.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2015-07-22 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2025-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Townsend, MD, Principal Investigator — University of Pennsylvania; David Kandzari, MD, Principal Investigator — Piedmont Hospital; Michael Böhm, MD, Principal Investigator — Universitätskliniken des Saarlandes; Kazuomi Kario, MD, Principal Investigator — Jichi Medical University
Locations (56):
- United States (32):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Stanford Hospital and Clinics, Stanford, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Memorial Hospital Jacksonville, Jacksonville, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Heart Institute, Atlanta, Georgia
  - Iowa Heart Center, West Des Moines, Iowa
  - University of Kentucky, Lexington, Kentucky
  - St Joseph Mercy Oakland, Pontiac, Michigan
  - Providence Hospital, Southfield, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Cardiology Associates Research LLC, Tupelo, Mississippi
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - North Shore University Hospital, Manhasset, New York
  - Weill Cornell Medical College/The New York Presbyterian Hospital, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Oregon Health & Science University Hospital, Portland, Oregon
  - PinnacleHealth Cardiovascular Institute, Harrisburg, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - AnMed Health, Anderson, South Carolina
  - Centennial Medical Center, Nashville, Tennessee
  - Baylor Heart & Vascular Hospital, Dallas, Texas
  - Charleston Area Medical Center, Charleston, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (3):
  - Alfred Hospital, Melbourne, Victoria
  - St. George Hospital, Kogarah
  - Royal Perth, Perth
- Klinikum Wels-Grieskirchen, Wels, Austria
- Canada (2):
  - Hamilton Heath, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
- Clinique Pasteur, Toulouse, France
- Germany (5):
  - Universitäts-Herzzentrum Freiburg - Bad Krozingen GmbH, Bad Krozingen
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum des Saarlandes, Homburg
  - Herzzentrum Leipzig, Universitätsklinik, Leipzig
  - Sana Kliniken Lübeck, Lübeck
- Greece (2):
  - Hippokration General Hospital of Athens, Athens
  - University General Hospital of Thessaloniki (AHEPA), Thessaloniki
- Galway University Hospital, Galway, Ireland
- Japan (5):
  - Higashi Takarazuka Satoh Hospital, Takarazuka, Hyōgo
  - Shonan Kamakura General Hospital, Kamakura, Okamoto
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Mitsui Memorial Hospital, Chiyoda City, Tokyo
  - Saiseikai Nakatsu Hospital, Osaka
- United Kingdom (4):
  - Royal Bournemouth Hospital, Bournemouth
  - Cardiff and Vale University Health Board - University Hospital of Wales, Cardiff
  - Royal Devon & Exeter NHS Foundation Trust, Exeter
  - Imperial College Healthcare NHS Trust, London

REFERENCES:
- [Derived] Kandzari DE, Mahfoud F, Townsend RR, Kario K, Weber MA, Schmieder RE, Tsioufis K, Pocock S, Liu M, DeBruin V, Brar S, Bohm M. Long-Term Safety and Efficacy of Renal Denervation: 24-Month Results From the SPYRAL HTN-ON MED Trial. Circ Cardiovasc Interv. 2025 Jul;18(7):e015194. doi: 10.1161/CIRCINTERVENTIONS.125.015194. Epub 2025 May 20. PMID 40391448
- [Derived] Townsend RR, Ferdinand KC, Kandzari DE, Kario K, Mahfoud F, Weber MA, Schmieder RE, Pocock S, Tsioufis K, David S, Steigerwalt S, Walton A, Hopper I, Bertolet B, Sharif F, Fengler K, Fahy M, Hettrick DA, Brar S, Bohm M. Impact of Antihypertensive Medication Changes After Renal Denervation Among Different Patient Groups: SPYRAL HTN-ON MED. Hypertension. 2024 May;81(5):1095-1105. doi: 10.1161/HYPERTENSIONAHA.123.22251. Epub 2024 Feb 5. PMID 38314554
- [Derived] Kandzari DE, Townsend RR, Kario K, Mahfoud F, Weber MA, Schmieder RE, Pocock S, Tsioufis K, Konstantinidis D, Choi J, East C, Lauder L, Cohen DL, Kobayashi T, Schmid A, Lee DP, Ma A, Weil J, Agdirlioglu T, Schlaich MP, Shetty S, Devireddy CM, Lea J, Aoki J, Sharp ASP, Anderson R, Fahy M, DeBruin V, Brar S, Bohm M; SPYRAL HTN-ON MED Investigators. Safety and Efficacy of Renal Denervation in Patients Taking Antihypertensive Medications. J Am Coll Cardiol. 2023 Nov 7;82(19):1809-1823. doi: 10.1016/j.jacc.2023.08.045. PMID 37914510
- [Derived] Mahfoud F, Kandzari DE, Kario K, Townsend RR, Weber MA, Schmieder RE, Tsioufis K, Pocock S, Dimitriadis K, Choi JW, East C, D'Souza R, Sharp ASP, Ewen S, Walton A, Hopper I, Brar S, McKenna P, Fahy M, Bohm M. Long-term efficacy and safety of renal denervation in the presence of antihypertensive drugs (SPYRAL HTN-ON MED): a randomised, sham-controlled trial. Lancet. 2022 Apr 9;399(10333):1401-1410. doi: 10.1016/S0140-6736(22)00455-X. Epub 2022 Apr 4. PMID 35390320
- [Derived] Kandzari DE, Hickey GL, Pocock SJ, Weber MA, Bohm M, Cohen SA, Fahy M, Lamberti G, Mahfoud F. Prioritised endpoints for device-based hypertension trials: the win ratio methodology. EuroIntervention. 2021 Apr 2;16(18):e1496-e1502. doi: 10.4244/EIJ-D-20-01090. PMID 33226002
- [Derived] Kario K, Weber MA, Bohm M, Townsend RR, Mahfoud F, Schmieder RE, Tsioufis K, Cohen SA, Fahy M, Kandzari DE. Effect of renal denervation in attenuating the stress of morning surge in blood pressure: post-hoc analysis from the SPYRAL HTN-ON MED trial. Clin Res Cardiol. 2021 May;110(5):725-731. doi: 10.1007/s00392-020-01718-6. Epub 2020 Aug 1. PMID 32740754
- [Derived] Bohm M, Townsend RR, Kario K, Kandzari D, Mahfoud F, Weber MA, Schmieder RE, Tsioufis K, Hickey GL, Fahy M, DeBruin V, Brar S, Pocock S. Rationale and design of two randomized sham-controlled trials of catheter-based renal denervation in subjects with uncontrolled hypertension in the absence (SPYRAL HTN-OFF MED Pivotal) and presence (SPYRAL HTN-ON MED Expansion) of antihypertensive medications: a novel approach using Bayesian design. Clin Res Cardiol. 2020 Mar;109(3):289-302. doi: 10.1007/s00392-020-01595-z. Epub 2020 Feb 7. PMID 32034481
- [Derived] Kandzari DE, Bohm M, Mahfoud F, Townsend RR, Weber MA, Pocock S, Tsioufis K, Tousoulis D, Choi JW, East C, Brar S, Cohen SA, Fahy M, Pilcher G, Kario K; SPYRAL HTN-ON MED Trial Investigators. Effect of renal denervation on blood pressure in the presence of antihypertensive drugs: 6-month efficacy and safety results from the SPYRAL HTN-ON MED proof-of-concept randomised trial. Lancet. 2018 Jun 9;391(10137):2346-2355. doi: 10.1016/S0140-6736(18)30951-6. Epub 2018 May 23. PMID 29803589
- [Derived] Kandzari DE, Kario K, Mahfoud F, Cohen SA, Pilcher G, Pocock S, Townsend R, Weber MA, Bohm M. The SPYRAL HTN Global Clinical Trial Program: Rationale and design for studies of renal denervation in the absence (SPYRAL HTN OFF-MED) and presence (SPYRAL HTN ON-MED) of antihypertensive medications. Am Heart J. 2016 Jan;171(1):82-91. doi: 10.1016/j.ahj.2015.08.021. Epub 2015 Sep 11. PMID 26699604

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Renal Denervation | Sham Procedure
Started | 206 | 131
Completed | 115 | 73
Not Completed | 91 | 58

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Renal Denervation | Sham Procedure | Total
Number analyzed (Participants) | 206 | 131 | 337
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.2 (9.0) | 54.6 (9.4) | 54.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 28 | 67
  Male | 167 | 103 | 270
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 17 | 10 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 25 | 60
  White | 71 | 48 | 119
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 81 | 48 | 129
Length of hypertension diagnosis [Count of Participants; unit: Participants]
  0-5 years | 62 | 24 | 86
  6-10 years | 37 | 27 | 64
  >10 years | 107 | 80 | 187
Office Blood Pressure [Mean (Standard Deviation); unit: mm Hg]
  Office Systolic Blood Pressure | 163.0 (7.7) | 163.1 (7.9) | 163.05 (7.8)
  Office Diastolic Blood Pressure | 101.2 (7.0) | 101.5 (7.3) | 101.4 (7.2)
24- hour Ambulatory Blood Pressure [Mean (Standard Deviation); unit: mm Hg]
  24- hour Ambulatory Systolic Blood Pressure | 149.6 (7.0) | 149.3 (7.0) | 149.5 (7.0)
  24-hour Ambulatory Diastolic Blood Pressure | 96.6 (7.6) | 95.7 (7.7) | 96.2 (7.65)

OUTCOME MEASURES:

1. Primary Outcome: Acute and Chronic Safety by Evaluating Incidence of Major Adverse Events
Description: The primary safety endpoint of the study is the incidence of Major Adverse Events (MAE), defined as a composite of the following events: All-cause mortality, End Stage Renal Disease (ESRD), Significant embolic event resulting in end-organ damage, Renal artery perforation requiring intervention, Renal artery dissection requiring intervention, Vascular complications, Hospitalization for hypertensive crisis not related to confirmed non-adherence with medications or the protocol, New renal artery stenosis >70%, confirmed by angiography and as a determined by the angiographic core laboratory, through one-month post-randomization (6- months for new renal artery stenosis).
Time Frame: From baseline to 1 month post-procedure (6 months for new renal artery stenosis)
Population: All randomized subjects are analyzed according to their randomized treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 206 | 131
Participants
  No MAE | 204 | 130
  Vascular Complication requiring intervention | 2 | 1

2. Primary Outcome: Change in Systolic Blood Pressure as Measured by 24-hour Ambulatory Blood Pressure Monitoring (ABPM)
Description: Baseline adjusted change (using Analysis of Covariance) in systolic blood pressure (SBP) from baseline (Screening Visit 2) to 6 months post-procedure as measured by 24-hour Ambulatory Blood Pressure Monitoring (ABPM).
Time Frame: From baseline to 6 months post-procedure
Population: All randomized subjects are analyzed according to their randomized treatment. Subjects who met the anti-hypertensive medication escape criteria (Office SBP>180 or <115 mmHg associated with symptoms of hypotension or safety concern requiring medication changes) are analyzed using Last Observation Carried Forward (LOCF) for their blood pressure measurements out to 6-months.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 192 | 116
mm Hg | -6.5 (10.7) | -4.5 (10.3)
Statistical Analysis 1: Comparison: Renal Denervation vs Sham Procedure; Test type: Superiority; p = 0.1194, ANCOVA — p<0.05 required for significance

3. Secondary Outcome: Change in Office Systolic Blood Pressure
Description: Change in office systolic blood pressure from baseline (Screening Visit 2) to 6 months post-procedure
Time Frame: From baseline to 6 months post-procedure
Population: Valid readings at time of data collection
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 199 | 126
mmHg | -9.9 (13.9) | -5.1 (13.2)

4. Secondary Outcome: Antihypertensive Medication Usage and Changes to 6-months
Description: Number of medications from baseline (Screening Visit 2) through 6 Months post-procedure
Time Frame: From baseline to 6-month post-procedure
Population: Prescribed daily medication reported
Measure: Mean (Standard Deviation); unit: Number of Daily Medications
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 206 | 131
Number of Daily Medications
  Baseline | 1.9 (.8) | 1.9 (0.8)
  6 Months: number analyzed (Participants) | 204 | 130
  6 Months | 1.9 (0.9) | 2.1 (0.9)

5. Secondary Outcome: Antihypertensive Medication Burden to 6-months
Description: Based on the prescribed medications reported, medication burden was calculated using Medication Index 2 score which is a composite index based on the doses of antihypertensive medications multiplied by the number of medications prescribed; all classes (ACE/ARB, calcium channel blockers, etc.) were considered equivalent in potency. Higher score indicates higher dosages being prescribed over the standard dose.
  Minimum value 0; No Maximum value
Time Frame: From baseline to 6 Months post-procedure
Population: Prescribed medications reported
Measure: Mean (Standard Deviation); unit: Medication Index 2 Score
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 206 | 131
Medication Index 2 Score
  Baseline | 2.8 (2.5) | 3.0 (2.6)
  6 Months: number analyzed (Participants) | 204 | 130
  6 Months | 2.9 (2.7) | 3.5 (3.2)

6. Secondary Outcome: Medication Changes
Description: Patients who had medication changes based on Medication Index 2 drug testing data. Medication Index 2 score is a composite index based on the doses of antihypertensive medications multiplied by the number of medications prescribed; all classes (ACE/ARB, calcium channel blockers, etc.) were considered equivalent in potency.
Time Frame: Baseline to 6-months post-procedure
Population: Confirmed via Drug Testing Data at both Baseline (Screening Visit 2) and 6-months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 200 | 128
Participants
  Increase | 37 | 35
  No Change | 131 | 80
  Decrease | 32 | 13

7. Secondary Outcome: Incidence of Achieving Target Office Systolic Blood Pressure
Description: Incidence of achieving target office systolic blood pressure (SBP<140 mmHg) at 6 months post- procedure.
Time Frame: From baseline to 6 months post-procedure
Population: Valid readings at time of data collection
Measure: Count of Participants; unit: Participants
Arm/Group | Renal Denervation | Sham Procedure
Number analyzed (Participants) | 199 | 126
Participants | 39 | 8

ADVERSE EVENTS:
Time Frame: Adverse Events through 6 months
Arm/Group | Renal Denervation | Sham Procedure
All-Cause Mortality (participants affected / at risk) | 0/206 | 0/131
Serious Adverse Events (participants affected / at risk) | 18/206 | 15/131
Other Adverse Events (participants affected / at risk) | 129/206 | 89/131
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Renal Denervation (N=206) | Sham Procedure (N=131)
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Atrial Flutter (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Adrenal Mass (Endocrine disorders) | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1 — General Disorders And Administration Site Conditions
Chest Discomfort (General disorders) | 0 | 1 — General Disorders And Administration Site Conditions
Non-Cardiac Chest Pain (General disorders) | 1 | 1 — General Disorders And Administration Site Conditions
Oedema Peripheral (General disorders) | 0 | 1 — General Disorders And Administration Site Conditions
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Vestibular Neuronitis (Infections and infestations) | 1 | 0
Viral Sepsis (Infections and infestations) | 1 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular Access Site Haematoma (Injury, poisoning and procedural complications) | 1 | 0
Vascular Access Site Pseudoaneurysm (Injury, poisoning and procedural complications) | 2 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Anogenital Warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Bladder Neck Obstruction (Renal and urinary disorders) | 0 | 1
Removal Of Foreign Body (Surgical and medical procedures) | 1 | 0
Raynaud's Phenomenon (Vascular disorders) | 1 | 0
Angina Unstable (Cardiac disorders) | 0 | 0
Retinal Detachment (Eye disorders) | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0
Chest Pain (General disorders) | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0
Simple Partial Seizures (Nervous system disorders) | 0 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 0
Syncope (Nervous system disorders) | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0
Renal Artery Stenosis (Renal and urinary disorders) | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Hypertensive Crisis (Vascular disorders) | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Renal Denervation (N=206) | Sham Procedure (N=131)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 2 | 2
Atrial Flutter (Cardiac disorders) | 1 | 0
Atrioventricular Block Second Degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 3 | 1
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Left Ventricular Failure (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Adrenal Mass (Endocrine disorders) | 1 | 0
Basedow's Disease (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 2
Primary Hyperaldosteronism (Endocrine disorders) | 1 | 0
Conjunctivitis Allergic (Eye disorders) | 1 | 0
Swelling Of Eyelid (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 0 | 1
Visual Impairment (Eye disorders) | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 3 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis Ulcerative (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Food Poisoning (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 1 | 0
Lip Swelling (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 0
Toothache (Gastrointestinal disorders) | 2 | 2
Adverse Drug Reaction (General disorders) | 1 | 1 — General Disorders And Administration Site Conditions
Asthenia (General disorders) | 1 | 1 — General Disorders And Administration Site Conditions
Chest Discomfort (General disorders) | 1 | 1 — General Disorders And Administration Site Conditions
Chest Pain (General disorders) | 1 | 4 — General Disorders And Administration Site Conditions
Cyst (General disorders) | 0 | 1 — General Disorders And Administration Site Conditions
Drug Intolerance (General disorders) | 1 | 0 — General Disorders And Administration Site Conditions
Fat Necrosis (General disorders) | 0 | 1 — General Disorders And Administration Site Conditions
Fatigue (General disorders) | 2 | 1 — General Disorders And Administration Site Conditions
Influenza Like Illness (General disorders) | 0 | 1 — General Disorders And Administration Site Conditions
Non-Cardiac Chest Pain (General disorders) | 1 | 1 — General Disorders And Administration Site Conditions
Oedema Peripheral (General disorders) | 6 | 12 — General Disorders And Administration Site Conditions
Peripheral Swelling (General disorders) | 3 | 2 — General Disorders And Administration Site Conditions
Puncture Site Haematoma (General disorders) | 1 | 0 — General Disorders And Administration Site Conditions
Pyrexia (General disorders) | 1 | 0 — General Disorders And Administration Site Conditions
Swelling (General disorders) | 0 | 1 — General Disorders And Administration Site Conditions
Vessel Puncture Site Haematoma (General disorders) | 1 | 0 — General Disorders And Administration Site Conditions
Vessel Puncture Site Induration (General disorders) | 1 | 0 — General Disorders And Administration Site Conditions
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Hepatic Lesion (Hepatobiliary disorders) | 1 | 0
Hepatic Steatosis (Hepatobiliary disorders) | 0 | 1
Contrast Media Reaction (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Bacterial Vaginosis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 0
Bursitis Infective (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Conjunctivitis Viral (Infections and infestations) | 1 | 0
Covid-19 (Infections and infestations) | 5 | 3
Cystitis (Infections and infestations) | 1 | 1
Eye Infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Fungal Foot Infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Gastrointestinal Viral Infection (Infections and infestations) | 0 | 1
Groin Abscess (Infections and infestations) | 1 | 0
Infectious Mononucleosis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 6
Localised Infection (Infections and infestations) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Ludwig Angina (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 2
Onychomycosis (Infections and infestations) | 0 | 1
Oral Herpes (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Pulpitis Dental (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 1
Rhinitis (Infections and infestations) | 0 | 1
Scrotal Abscess (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 1
Tinea Cruris (Infections and infestations) | 0 | 1
Tinea Pedis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 1
Tooth Abscess (Infections and infestations) | 1 | 0
Tooth Infection (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 3
Urethritis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 2
Vestibular Neuronitis (Infections and infestations) | 1 | 0
Viral Sepsis (Infections and infestations) | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1
Wound Infection Staphylococcal (Infections and infestations) | 1 | 0
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Exposure To Extreme Temperature (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 1 | 0
Incision Site Complication (Injury, poisoning and procedural complications) | 1 | 0
Incision Site Pain (Injury, poisoning and procedural complications) | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Meniscus Injury (Injury, poisoning and procedural complications) | 1 | 0
Muscle Strain (Injury, poisoning and procedural complications) | 0 | 1
Post Procedural Discomfort (Injury, poisoning and procedural complications) | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 1
Skin Abrasion (Injury, poisoning and procedural complications) | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 2 | 0
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 | 0
Stoma Prolapse (Injury, poisoning and procedural complications) | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1
Tooth Fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 | 0
Vaccination Complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular Access Site Bruising (Injury, poisoning and procedural complications) | 2 | 0
Vascular Access Site Haematoma (Injury, poisoning and procedural complications) | 10 | 10
Vascular Access Site Haemorrhage (Injury, poisoning and procedural complications) | 2 | 1
Vascular Access Site Pain (Injury, poisoning and procedural complications) | 5 | 0
Vascular Access Site Pseudoaneurysm (Injury, poisoning and procedural complications) | 2 | 1
Vascular Access Site Thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Wound Secretion (Injury, poisoning and procedural complications) | 1 | 0
Blood Cholesterol Increased (Investigations) | 1 | 0
Blood Creatinine Increased (Investigations) | 1 | 3
Blood Glucose Increased (Investigations) | 1 | 0
Blood Potassium Decreased (Investigations) | 2 | 0
Blood Potassium Increased (Investigations) | 0 | 1
Blood Pressure Abnormal (Investigations) | 1 | 0
Blood Pressure Increased (Investigations) | 6 | 4
Blood Pressure Orthostatic Decreased (Investigations) | 0 | 1
Blood Uric Acid Increased (Investigations) | 1 | 0
C-Reactive Protein Increased (Investigations) | 0 | 1
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 1
Glycosylated Haemoglobin Increased (Investigations) | 1 | 1
Heart Rate Increased (Investigations) | 1 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 0
Lipids Increased (Investigations) | 1 | 0
Liver Function Test Increased (Investigations) | 1 | 1
Oxygen Saturation Decreased (Investigations) | 1 | 0
Pancreatic Enzymes Increased (Investigations) | 1 | 0
Renal Function Test Abnormal (Investigations) | 1 | 0
Troponin T Increased (Investigations) | 0 | 1
Weight Increased (Investigations) | 0 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 1 | 1
Gout (Metabolism and nutrition disorders) | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 8
Hypolipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 12 | 4
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Facet Joint Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Inguinal Mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 2 | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 4 | 2
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 | 5
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases To Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carpal Tunnel Syndrome (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 5 | 6
Dizziness Postural (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 7 | 9
Hypoaesthesia (Nervous system disorders) | 0 | 2
Ischaemic Stroke (Nervous system disorders) | 0 | 1
Lethargy (Nervous system disorders) | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 2
Nerve Compression (Nervous system disorders) | 1 | 0
Neuropathy Peripheral (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 3 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Sciatic Nerve Neuropathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 2
Anxiety (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 1 | 0
Mental Disorder (Psychiatric disorders) | 1 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 1
Neuropsychiatric Symptoms (Psychiatric disorders) | 0 | 1
Poor Quality Sleep (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Bladder Neck Obstruction (Renal and urinary disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Hypertonic Bladder (Renal and urinary disorders) | 0 | 1
Micturition Urgency (Renal and urinary disorders) | 0 | 1
Renal Artery Dissection (Renal and urinary disorders) | 2 | 0
Renal Cyst (Renal and urinary disorders) | 3 | 0
Urinary Incontinence (Renal and urinary disorders) | 0 | 1
Urinary Retention (Renal and urinary disorders) | 0 | 1
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 1
Breast Mass (Reproductive system and breast disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Scrotal Cyst (Reproductive system and breast disorders) | 0 | 1
Testicular Pain (Reproductive system and breast disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Cough Variant Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Respiratory Depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 2
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Swelling (Skin and subcutaneous tissue disorders) | 0 | 1
Transient Acantholytic Dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Removal Of Foreign Body (Surgical and medical procedures) | 1 | 0
Wisdom Teeth Removal (Surgical and medical procedures) | 0 | 1
Arterial Spasm (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 6
Hypertensive Crisis (Vascular disorders) | 0 | 1
Hypertensive Urgency (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 2 | 1
Iliac Artery Dissection (Vascular disorders) | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 1
Raynaud's Phenomenon (Vascular disorders) | 1 | 0
Vasospasm (Vascular disorders) | 1 | 0
Anogenital Warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Angina Unstable (Cardiac disorders) | 0 | 0
Cardiac Hypertrophy (Cardiac disorders) | 0 | 0
Liddle's Syndrome (Congenital, familial and genetic disorders) | 0 | 0
Retinal Detachment (Eye disorders) | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0
Paraesthesia Oral (Gastrointestinal disorders) | 0 | 0
Stomach Mass (Gastrointestinal disorders) | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0
Pain (General disorders) | 0 | 0 — General Disorders And Administration Site Conditions
Acute Sinusitis (Infections and infestations) | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0
Ear Infection (Infections and infestations) | 0 | 0
Gastrointestinal Infection (Infections and infestations) | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0
Bone Contusion (Injury, poisoning and procedural complications) | 0 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 0
Subcutaneous Haematoma (Injury, poisoning and procedural complications) | 0 | 0
Aortic Bruit (Investigations) | 0 | 0
Liver Function Test Abnormal (Investigations) | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 | 0
Bladder Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0
Bell's Palsy (Nervous system disorders) | 0 | 0
Cognitive Disorder (Nervous system disorders) | 0 | 0
Exertional Headache (Nervous system disorders) | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0
Simple Partial Seizures (Nervous system disorders) | 0 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0
Cystitis Noninfective (Renal and urinary disorders) | 0 | 0
Renal Artery Stenosis (Renal and urinary disorders) | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT02439775/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT02439775/SAP_001.pdf